CLINICAL TRIAL: NCT06856603
Title: OLIGO-10: Stereotactic Ablative Radiation Therapy for Metastatic Patients (6-10 Metastases): A Prospective Phase II Single-Arm Trial
Brief Title: OLIGO-10: Stereotactic Ablative Radiation Therapy for Metastatic Patients With 6 to 10 Metastatic Sites
Acronym: OLIGO-10
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Konstantin Gordon, Principal Investigator, National Medical Research Radiological Centre of the Ministry of Health of Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024_06_13
Record Dates: First submitted 2025-02-12; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Disease
Keywords: Metastatic Disease; Stereotactic radiation therapy; Stereotactic body radiation therapy; Stereotactic ablative radiation therapy; Oligometastatic Disease
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: SABR for Extra- and Intracranial Metastatic Disease with 6-10 Sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-arm: Stereotactic Ablative Radiotherapy (SABR) for 6-10 mts (Other): The method of stereotactic ablative radiation therapy will be used in patients with metastatic tumors (6-10 sites) of various localizations, following the current line of chemotherapy (T1-4, N0-3, M0-1), and who are over 18 years old at the time of treatment initiation.
  Interventions: Radiation: stereotactic radiation therapy in ablative doses to each metastatic site

INTERVENTIONS:
Radiation: stereotactic radiation therapy in ablative doses to each metastatic site — Stereotactic ablative radiation therapy will be utilized for each metastatic site in patients with 6 to 10 sites of metastasis (persistent or progressive disease).

SUMMARY:
Currently, the standard of care for patients with diagnosed metastatic cancer is drug therapy (chemotherapy, targeted therapy, or immunotherapy). However, the approach to oligometastatic disease (1-5 metastases) is evolving. An increasing number of de novo, persistent, and progressive oligometastatic tumors are now being treated with curative intent, with radiation therapy among the most effective treatment options, applied to metastatic sites in ablative doses. Emerging results from the SABR-COMET 3 and 5 trials, which investigate stereotactic ablative radiotherapy for patients with 1-3 and 1-5 metastatic sites, demonstrate a clear improvement in overall survival. However, patients with more than five metastases remain in a gray area.

The aim of our study is to assess the safety and effectiveness of radiation treatment for patients with tumors of various localizations and 6 to 10 metastases in the bones and internal organs. Stereotactic radiation therapy will be applied to patients with persistent or progressive metastatic forms of tumors, without changing their ongoing drug therapy regimen.

DETAILED DESCRIPTION:
1. A patient with a previously verified diagnosis of a malignant neoplasm of any localization (ICD 10-11 codes C) who meets the inclusion criteria, after approval by the tumor board for the study group, will undergo the following procedures:

   Three-dimensional/four-dimensional computed tomography for simulation using specialized fixation devices (the choice of the CT method and fixation devices will depend on the location of the metastasis).

   The resulting images will be added to the contouring program.

   Delineation of targets and organs at risk will be performed.

   Clinical volumes and error margins will be determined.
2. The total dose per target and dose limits for critical structures will be prescribed.

   Dosimetric planning for the course of external beam radiation therapy will be carried out.

   Irradiation sessions will be conducted on a linear accelerator with a multi-leaf collimator, including a function for visual control of the target using cone beam tomography with kilo-voltage/mega-voltage radiation.

   When the target is localized in the lungs, liver, or adrenal glands, to reduce the radiation load on surrounding healthy tissues and achieve necessary control over the position of the metastasis, irradiation will be performed with a deep breath hold or at specific phases of respiration.
3. Tumor Localization / Description / Total Focal Dose (Gy) / Number of Fractions / Single Focal Dose (Gy) / Irradiation Mode:

   Lung Tumors:

   Tumors ≤ 3 cm located in the parenchyma: TD 45 Gy in 3 fractions with 15 Gy each day Tumors adjacent to the chest wall or < 3 cm: TD 50 Gy in 5 fractions with 10 Gy each day Tumors within 2 cm of the mediastinum or brachial plexus: TD 60 Gy in 8 fractions with 7.5 Gy each day Bones: TD 24 Gy in 3 fractions with 8 Gy each day

   Brain Metastases:

   Tumor volume from 0.5 to 5 cm³: TD 20-22 Gy in 1 fraction at a time Tumor volume from 5 to 10 cm³: TD 16-18 Gy or TD 18-20 Gy in 1 fraction at a time Liver: Radiation regimen selection based on the tolerance of surrounding tissues and proximity to critical structures: TD 30-60 Gy in 3-8 fractions with 6-15 Gy each day

   Adrenal Glands: TD 60 Gy in 8 fractions with 7.5 Gy each day
4. Expected Duration of Patient Participation in Clinical Testing:

Pre-hospital period: Comprehensive examination of the patient before treatment. Inpatient period: Includes pre-radiation preparation for up to 3 working days, SABR treatment for 1 to 8 working days.

Follow-up period: 3, 6, 9, and 12 months post-treatment; thereafter, follow-up will occur every 6 months up to 60 months.

Collection and processing of received data.

ELIGIBILITY:
Inclusion Criteria:

* ECOG status 0-3
* Persistent or progressive cancer disease with 6 to 10 metastases
* ≤ 5 metastases in one organ
* Life expectancy > 6 months for intracranial lesions
* Inability to surgically resect all metastatic lesions
* Positive tumor board decision for trial inclusion
* Signed informed consent

Exclusion Criteria:

* ECOG status 4
* De novo metastatic disease
* Radiological complete response after drug therapy
* Brain metastasis only
* Brain metastasis > 3 cm, requiring neurosurgery
* Size of any metastasis > 5 cm
* Previous radiation therapy for any metastatic site
* Leptomeningeal, pleural, or peritoneal carcinomatosis
* Spinal cord compression, requiring neurosurgery
* Invasion of great vessels, skin, or GI tract
* Negative tumor board decision for trial inclusion
* Unsigned informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment safety | End of years 1, 2, 3, 4, 5 (study completion)
  Radiation-induced toxicity (type and corresponding grade 1 to 5) will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 scale.

SECONDARY OUTCOMES:
Effectiveness (PFS) | From the date of initiation until the date of documented disease progression, assessed over a period of up to 60 months.
  Progression-free survival, assessed in months
Effectiveness (LC) | From the date of initiation until the date of documented radiological signs of metastasis relapse, assessed over a period of up to 60 months.
  Local control for irradiated metastatic sites, assessed in months
Effectiveness (OS) | From the date of initiation until the date of death from any cause, assessed over a period of up to 60 months.
  Overall survival, assessed in months
Time-to-CTX-change | End of years 1, 2, 3, 4, 5 (study completion)
  Period of current drug line prolongation, assessed in months

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Kaprin, PhD, Study Chair — National Medical Research Radiological Centre of the Ministry of Health of Russia
Locations (1):
- A. Tsyb Medical Radiological Research Center, Obninsk, Kaluga Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request from the principal investigator for researchers, who meet the criteria for access to confidential data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: unlimited
Access Criteria: informed consent for personal data non-disclosure